CLINICAL TRIAL: NCT06784479
Title: A Randomized Clinical Trial to Evaluate the Sedative Effect of the Combination of Remimazolam and Propofol in Drug-induced Sleep Endoscopy
Brief Title: Combination of Remimazolam and Propofol During Drug-induced Sleep Endoscopy
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Dan Liu (Other)
Responsible Party: Sponsor-Investigator, Dan Liu, Master of Medicine, attending physician, Tianjin Medical University General Hospital
Organization: Tianjin Medical University General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: IRB2024-YX-607-01; 82300120 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2024-12-31; First posted 2025-01-20 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Sedative Effect During Drug-induced Sleep Endoscopy; Obstructive Sleep Apnea (OSA)
Keywords: drug-induced sleep endoscopy; remimazolam; propofol; Obstructive sleep apnea; airway collapsibility
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — remimazolam; Propofol; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Application of remimazolam and propofol to achieve satisfactory sedative effect (Experimental)
  Interventions: Drug: Remimazolam and Propofol
- Application of propofol to achieve satisfactory sedative effect (Active Comparator)
  Interventions: Drug: Propofol
- Application of midazolam and propofol to achieve satisfactory sedative effect (Active Comparator)
  Interventions: Drug: Midazolam and propofol

INTERVENTIONS:
Drug: Remimazolam and Propofol — Application of Remimazolam and Propofol to induce sleep
  Arms: Application of remimazolam and propofol to achieve satisfactory sedative effect
Drug: Propofol — Application of Propofol to induce sleep
  Arms: Application of propofol to achieve satisfactory sedative effect
Drug: Midazolam and propofol — Application of Midazolam and Propofol to induce sleep
  Arms: Application of midazolam and propofol to achieve satisfactory sedative effect

SUMMARY:
This study helps patients find the optimal sedation regimen in drug-induced sleep endoscopy

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with sleep apnea hypopnea syndrome were included

Exclusion Criteria:

* Patients were excluded if they had nasal obstruction, significantly deviated nasal septum, nasal turbinate hypertrophy, or nasal polyps. Patients with uncontrolled heart failure, renal insufficiency, diabetes, or hyperthyroidism were also excluded. Patients were also excluded if taking medications that could affect upper airway muscle function, such as ben- zodiazepines and muscle relaxants.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Sedative effect-Adequate sedation time | During procedure (From the start of medication to adequate sedation time), an average of 5min
  The doctor evaluate the time it takes for the patient to reach a state of sufficient sedation
Sedative effect-operation time | From the start of drug induced sleep endoscopy to the complete the operation, an average of 10min
  Adequate sedation time, hemodynamic response, operation time, sedation to recovery time, wake-up time
Sedative effect-sedation to recovery time | The time period of the end of operation to complete wakefulness,through operation completion, an average of 30min
  The process of a patient recovering from anesthesia to complete wakefulness
Sedative effect-sedation to wake-up time | During procedure (The time period of the doctor's call to the patient's awakening from anesthesia), an average of 10min
  The process of the patient wakes up from anesthesia

SECONDARY OUTCOMES:
Procedure-related adverse effect-The need for antidote administration | During procedure (From the start of drug induced sleep endoscopy to the complete awakening of the patient)
  Percentage of patients need for antidote administration
Procedure-related adverse effect-The occurrence of tachycardia | During procedure (From the start of drug induced sleep endoscopy to the complete awakening of the patient)
  Percentage of patients affected tachycardia（ECG monitor）
Procedure-related adverse effect-The occurrence of hypotension | During procedure (From the start of drug induced sleep endoscopy to the complete awakening of the patient)
  Percentage of patients affected hypotension（ECG monitor）
Procedure-related adverse effect-The occurrence of hypoxemia | During procedure (From the start of drug induced sleep endoscopy to the complete awakening of the patient)
  Percentage of patients affected hypoxemia（ECG monitor）
The degree of patient and physician satisfaction | During procedure (the start of drug induced sleep endoscopy to the complete awakening of the patient)
  The percentage of patient and physician satisfacted with the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Respiratory Endoscopy Center of Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality, China